CLINICAL TRIAL: NCT01737190
Title: PEEP Guided by Esophageal Balloon Measurement and Its Effect on Recruitment Maneuver
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Soroksky Arie, Dr., Wolfson Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0161-12-WOMC
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: ARDS
Keywords: esophageal pressure; ARDSnet protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PEEP guided by Esophageal pressure + Recruitment maneuver. (Experimental): Upon patient recruitment Esophageal balloon will be inserted and esophageal / pleural pressure will be measured. Thereafter, Inspiratory pressures and PEEP will be adjusted according to well established criteria. Inspiratory pressure and PEEP will be adjusted to achieve the best lung compliance possible while not exceeding transpulmonary end Inspiratory pressure of 25 to 30 cm H2O, and at the same time maintaining a positive transpulmonary end expiarory pressure of not more than 5 cm H2O.
  A recruitment maneuver with application of 40 cm H2O for up to 40 seconds will be performed.
  Interventions: Other: PEEP guided by Esophageal pressure + Recruitment maneuver

INTERVENTIONS:
Other: PEEP guided by Esophageal pressure + Recruitment maneuver — Upon patient recruitment Esophageal balloon will be inserted and esophageal / pleural pressure will be measured. Thereafter, Inspiratory pressures and PEEP will be adjusted according to well established criteria. Inspiratory pressure and PEEP will be adjusted to achieve the best lung compliance possible while not exceeding transpulmonary end Inspiratory pressure of 25 to 30 cm H2O, and at the same time maintaining a positive transpulmonary end expiarory pressure of not more than 5 cm H2O.
  A recruitment maneuver with application of 40 cm H2O for up to 40 seconds will be performed.

SUMMARY:
The aim of the study is to examine the effects of two different levels of PEEP on subsequent standard recruitment maneuver.

DETAILED DESCRIPTION:
In this study we will examine the effects of two levels of PEEP on subsequent recruitment maneuver. In the first group a recruitment maneuver will be performed in patients who are ventilated with PEEP level set according to the ARDS network algorithm.

Patients will then be crossed over to a study arm where another recruitment maneuver will be performed while PEEP is adjusted according to esophageal pressure measurements.

ELIGIBILITY:
Inclusion Criteria:

20 Man and women older than 18 years will be recruited.

Patients with acute respiratory failure of any cause who are mechanically ventilated according to the ARDS network recommendations will be considered for inclusion to the study.

To be included in the study a prerequisite of high peak Inspiratory pressure (plateau pressure of 25 to 30 cmH2O) has to be present, and at least one of the following four severity inclusion criteria has to be met.

1 - Low Total Respiratory system compliance (CT), defined as less than 50ml/cmH2O. 2 - PaO2 /FIO2 ratio of less than 300. 3 - Need for a PEEP greater than 10 cmH2O to maintain SaO2 of > 90%. 4 - PCO2 over 60 mmHg, or PH less than 7.2 that is attributed to respiratory acidosis.

Exclusion Criteria:

Patients with any of the following will be excluded from the study. Previous lung or chest wall surgery, previous esophageal surgery, known Achalasia or any other esophageal motility or spasm disorder, presence of chest thoracostomy tube, and any significant chest wall abnormality such as kyphoskoliosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
oxygenation | 4 hours
  the primary end point in both groups will be oxygenation improvement after each intervention in each arm.

SECONDARY OUTCOMES:
lung compliance | 4 hours
  after each intervention lung compliance will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Arie Soroksky, M.D., Principal Investigator — Wolfson MC
Locations (1):
- E. Wolfson MC, Holon, Israel